CLINICAL TRIAL: NCT02541435
Title: Acute and Long-term Cardiovascular Toxicity After Modern Radiotherapy for Breast Cancer - a Prospective Longitudinal Study
Brief Title: Acute and Long-term Cardiovascular Toxicity After Modern Radiotherapy for Breast Cancer
Status: Recruiting | Type: Observational
Sponsor: St. Olavs Hospital (Other)
Collaborators: Norwegian University of Science and Technology (Other); Alesund Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2015/583
Record Dates: First submitted 2015-09-01; First posted 2015-09-04 (Estimated); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Breast Neoplasms; Cardiovascular Diseases
Keywords: Radiotherapy; Biological markers; Magnetic resonance imaging; Echocardiography; Tomography, X-Ray Computed; Risk factors; Heart; Quality of Life
MeSH Terms: conditions — Breast Neoplasms; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- conventional radiotherapy: 450 breast cancer patients treated with conventional radiotherapy with or without anthracyclines and/or trastuzumab during 2007-2012
- breath controlled radiotherapy: 350 breast cancer patients treated with laser assisted breath controlled radiotherapy with or without anthracyclines and/or trastuzumab during 2015-2017
- controls: per participating patient 2 age-matched female controls from the HUNT-3 population (total 800)

SUMMARY:
In Europe, breast cancer is by far the most common form of cancer diagnosed in women today, accounting for 29% of all cases. The 5-year survival rate is approximately 90%. Surgery is usually combined with radiotherapy (RT), anthracyclines, aromatase inhibitors and/or trastuzumab (Herceptin) which all have improved the life expectancy and survival in breast cancer patients.

Unfortunately, RT is associated with a broad spectrum of cardiovascular diseases, which includes coronary artery disease, valvular dysfunction, congestive heart failure and stroke, and is the most common non-malignancy cause of death. During the last two decades, RT regimens for breast cancer have changed and the doses of radiation to which the heart is exposed are now potentially lower due to new and improved RT techniques. However, there are no data on whether these new regimes decrease the risk of cardiovascular disease.

In this study the incidence and prevalence of cardiovascular diseases will be estimated 8 and 15 years after both conventional and laser assisted breath controlled RT, and compared with cardiovascular diseases in the general female population. A further aim is to evaluate signs and prevalence of acute cardiotoxicity from RT with the use of cardiac magnetic resonance imaging, coronary fractional flow reserve, ECG and inflammatory and cardiac biomarkers and to investigate whether these signs can predict later cardiovascular disease. The importance of traditional cardiovascular risk factors (age, hypertension, hypercholesterolemia, smoking habits and physical activity, as registered before RT) will also be evaluated.

DETAILED DESCRIPTION:
The study is an observational study. In 2007-2012 conventional RT was part of the common treatment regime for breast cancer, but has recently been replaced by laser assisted breath controlled RT. Thus, two cohorts of breast cancer patients treated with different modes of RT will be followed for the development of cardiovascular disease for the subsequent 15 years.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of breast cancer
* expected life-expectancy above 10 years

Exclusion Criteria:

* Not willing to participate

Ages: 30 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: women treated for breast cancer with radiotherapy
Sampling Method: Non-Probability Sample
Enrollment: 1600 (Estimated)
Dates: Start 2016-11 (Actual); Primary Completion 2029-12 (Estimated); Study Completion 2036-12 (Estimated)

PRIMARY OUTCOMES:
incidence of cardiovascular disease | 8 years
  compared with corresponding estimates from the female general population (HUNT-registry data, age-matched sample)
incidence of cardiovascular disease | 15 years
  compared with corresponding estimates from the female general population (HUNT-registry data, age-matched sample)

CONTACTS AND LOCATIONS:
Overall Officials: Jo-Åsmund Lund, md phd, Study Chair — St. Olavs Hospital
Locations (2):
- Norway (2):
  - Ålesund Hospital, Ålesund
  - St Olavs University Hospital, Trondheim

REFERENCES:
- [Background] Reidunsdatter RJ, Rannestad T, Frengen J, Frykholm G, Lundgren S. Early effects of contemporary breast radiation on health-related quality of life - predictors of radiotherapy-related fatigue. Acta Oncol. 2011 Nov;50(8):1175-82. doi: 10.3109/0284186X.2011.604345. Epub 2011 Aug 28. PMID 21871005